CLINICAL TRIAL: NCT05691673
Title: The Effect of Training Periodization on the Upper Extremity Force-velocity Profile in Swimmers During a Macro Cycle
Brief Title: Upper Extremity Force-velocity Profile in Swimmers
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ferhat Öztürk, Principal Investigator, Hacettepe University
Other Study IDs: GO 21/1151
Record Dates: First submitted 2022-12-16; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Upper Extremity Injury
Keywords: swimming; performance; strength; plyometric
MeSH Terms: conditions — Arm Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — Observational during 16 weeks

SUMMARY:
The aim of this study was to measure the changes in the upper extremity force-velocity profile of young swimmers at different training periods during a training season

DETAILED DESCRIPTION:
Tested at each experimental test time point (Baseline: E1, post-general preparation: E2, post-specific E3 and post-competition season: E4). To measure the upper extremity force-velocity parameters, the countermovement push-up test was performed using the force plate

ELIGIBILITY:
Inclusion Criteria:

* 15-18 age
* go to training regularly

Exclusion Criteria:

* upper extremity surgery in the last 1 year
* pain during the tests

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Health young swimmers in competitive club
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2022-08-19 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
The change in the parameters of the force (Newton) obtained from the force platform with countermovement push up from the baseline to the end of the season. | Baseline: E1, (week 0) post-general preparation: E2 (week 6), post-specific E3 ( week12) and post-competition season: E4 (week 16).
  Tested at each experimental test time point (Baseline: E1, post-general preparation: E2, post-specific E3 and post-competition season: E4). To measure the upper extremity force-velocity parameters, the countermovement push-up test was performed using the force plate.
velocity (m/s) | Baseline: E1, (week 0) post-general preparation: E2 (week 6), post-specific E3 ( week12) and post-competition season: E4 (week 16).
  Tested at each experimental test time point (Baseline: E1, post-general preparation: E2, post-specific E3 and post-competition season: E4). To measure the upper extremity force-velocity parameters, the countermovement push-up test was performed using the force plate.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Undecided